CLINICAL TRIAL: NCT05735535
Title: Multi-center Study to Evaluate Virological Efficacy, Safety Tolerability, Drug Exposure and Patients' Reported Outcomes Over 48 Weeks Following Randomization to 2-drug Therapy With DTG/3TC FDC or Continuing Current Antiretroviral Tenofovir (TAF or TDF)-Containing Regimen (T-CR) in HIV-1 Infected Virologically Suppressed
Brief Title: Women in Dual With Dolutegravir
Acronym: Woddol4455
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4455
Record Dates: First submitted 2023-02-01; First posted 2023-02-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Antiviral Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 3TC/DTG (Experimental): ·To evaluate efficacy of switching to a two-drug one-pill regimen with DTG/3TC
  Interventions: Drug: Antiviral Agents
- TDF Regimen (Active Comparator): comparision arm to maintaining the three-drugs regimen in women currently receiving any three-drug regimen containing Tenovofir (TAF or TDF) (e.g. TAF/F/E/C; TAF/F/RPV; TDF/F/RPV; TAF/F+PI/C; TAF/F+PI/r; TDF/F/PI/r; TAF/F+DTG; TDF/F/DTG; TAF/F+RTG; TDF/F/RTG; TAF/F/BIC) who are virologically suppressed.
  Interventions: Drug: Antiviral Agents

INTERVENTIONS:
Drug: Antiviral Agents — two-drug one-pill once day

SUMMARY:
Strategies for optimizing antiretroviral treatment in virologically suppressed patients are still a major challenge in the field of HIV. These strategies include improving the toxicity and tolerability of drugs in the short and long term, such as replacing toxic agents with safer ones or reducing the number of drugs in the combination. Tenofovir alafenamide (TAF) is a novel prodrug of tenofovir (TFV) that is converted intracellularly to the active form, resulting in higher concentrations of TFV diphosphate in circulating lymphocytes than those obtained with tenofovir disoproxil fumarate (TDF). Because of these pharmacokinetic properties, TAF results in 91% lower plasma exposure to TFV. Phase 3 studies have established the virological noninferiority of TAF to TDF, with a lower frequency of renal and bone adverse events. Replacing TDF with TAF may be a safe and effective option to reduce toxicities when switching from one ARV strategy to another and, to date, could represent the optimization of a three-drug regimen. Dolutegravir (DTG) is a potent INSTI that exhibits rapid and potent viral load reduction and a high barrier to resistance.

ELIGIBILITY:
Inclusion Criteria:

* Female individuals
* HIV-1 documented infection
* Age > 18 years
* Being on an effective (pVL < 50 copies/ml) three-drug cART regimen containing tenofovir (TAF or TDF) (e.g. TAF/F/E/C; TAF/F/RPV; TDF/F/RPV; TAF/F+PI/C; TDF/F/PI/c; TAF/F+PI/r; TDF/F/PI/r; TAF/F+DTG; TDF/F/DTG; TAF/F+RTG; TDF/F/RTG; TAF/F/BIC) for at least 3 months before the screening. Two consecutive HIV-1 RNA determinations below the determination threshold before enrollment are required
* No known allergy or intolerance to NRTIs, NNRTIs or INSTIs
* Women of childbearing potential will be required to adopt an effective birth control system throughout the study period
* Subjects able to comply with the protocol requirements
* Informed consent signed

Exclusion Criteria:

* Having failed virologically any previous ART regimen · Evidence of any 3TC (presence of M184V/I or K65R/E/N) or INSTI resistance · Having ever been treated with mono or dual ARV therapies subsequently intensified to three-drug cART regimen
* Pregnancy or breast-feeding or not willing to use effective contraception if they are of child bearing potential
* An active malignancy or OI requiring active treatment (prophylactic regimens are allowed) · HBV infection · A life expectancy < 2 years

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
HIV-RNA < 50 copies/ml | 96 weeks
  Proportion of patients maintaining a HIV-RNA < 50 copies/ml according to FDA snapshot algorithm at 48 weeks according to an ITT NC = failure approach in which all randomized patients will be included and considered failures independently of the reason they did not complete the follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione PoliclinicoAgostino Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No